CLINICAL TRIAL: NCT00136669
Title: Acupuncture For Pancreatic Cancer Pain: A Randomized Phase III Study
Brief Title: Acupuncture For Pancreatic Cancer Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 03-106
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2006-09-08 (Estimated); Status verified 2006-09

CONDITIONS: Pancreatic Neoplasms; Pain
Keywords: Acupuncture; Pain; Pancreatic Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms; Pain | interventions — Acupuncture Therapy

INTERVENTIONS:
Procedure: Acupuncture

SUMMARY:
Pain is a common problem in patients with pancreatic cancer. Some patients suffer from pain despite medication. We, the researchers at Memorial Sloan-Kettering Cancer Center, are conducting a Phase III study to determine the effects of acupuncture on pain in patients with pancreatic cancer. The purpose of a Phase III study is to determine whether or not a treatment is helpful. This study will include about 60 patients.

Acupuncture is the insertion of very fine needles into the skin to treat symptoms. In recent years, researchers have found evidence that acupuncture is useful in treating a variety of conditions, including headache, nausea, and pain.

DETAILED DESCRIPTION:
The main aim of this pancreatic cancer pain trial is to determine the effects of a single, practitioner-given acupuncture treatment followed by semi-permanent acupuncture studs. Our primary endpoint is subjective; therefore, a placebo control will be applied with patients blinded to treatment allocation.

In clinical practice, acupuncturists individualize treatment: two patients with a similar conventional diagnosis may receive different point prescriptions depending on the acupuncture differential diagnosis. Randomized trials of acupuncture can either prescribe a fixed treatment formula in terms of the number of sessions and points to be used, or allow practitioners to exercise clinical judgment in individualizing care. There has been considerable debate in the methodological literature about the merits of each approach. The use of a fixed treatment schedule increases the reproducibility of the findings but is said, by practitioners, to generally reduce treatment effectiveness. In this trial, we have developed an approach that allows practitioners to individualize treatments in a manner that allows exact replication, by specifying particular point locations to be used depending on the sites where a patient experiences pain. Point locations for this and for all of our acupuncture studies are determined by our licensed, credentialled acupuncturists.

Following accrual of the initial 10-15 patients, we will review treatment compliance, blinding and accrual. Adjustments will be made to deal with compliance issues, to facilitate placebo blinding, or deal with recruitment problems for the remainder of the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pancreatic adenocarcinoma.
* First baseline current pain score of 3 or above on a 0 - 10 numerical rating scale.
* In the opinion of the treating physician or a medically qualified investigator, the patient's pain syndrome is the result of underlying cancer.
* Patient OR caregiver must be willing and able to apply pressure to each point using small circular movements with the fingers twice per day.

Exclusion Criteria:

* Primary cause of pain is procedural (e.g. postoperative pain).
* Acupuncture treatment in the past six weeks. Patients should not receive acupuncture during the one week period of the study.
* Neutropenia defined as absolute neutrophil count (ANC) <1000/microliter.
* Cardiac conditions constituting high or moderate risk of endocarditis as defined by the American Heart Association criteria.
* Patient contraindicated for phlebotomy, as phlebotomy needles are much larger than acupuncture needles.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2003-09; Study Completion 2005-09

PRIMARY OUTCOMES:
To determine whether acupuncture reduces pain in pancreatic cancer patients more effectively than placebo
To determine the duration of acupuncture effects

CONTACTS AND LOCATIONS:
Overall Officials: Barrie R. Cassileth, Ph.D., Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: (Memorial Sloan-Kettering Cancer Center) — http://mskcc.org